CLINICAL TRIAL: NCT05475340
Title: Open Label Study for the Use of Transcranial Ultrasound Treatment of Tremor
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Neurological Associates of West Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fUS-Tremor
Record Dates: First submitted 2022-07-21; First posted 2022-07-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Tremor; Parkinson Disease; Essential Tremor
MeSH Terms: conditions — Tremor; Parkinson Disease; Essential Tremor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental (Experimental): Participants will undergo ten to thirty minutes of transcranial ultrasound treatment. The sanitation device will be aimed at the hypothalamus. Targeting will include reference to scalp fiducials based on the obtained MRI; confirmation of target accuracy will either be obtained by Doppler waveform confirmation or optical tracking technology which co-registers patient neuroimaging with real space.
  Interventions: Device: Focused Ultrasound

INTERVENTIONS:
Device: Focused Ultrasound — The DWL Doppler ultrasound device enables visual and auditory waveform confirmation of the middle cerebral artery, and optical tracking technology (e.g., AntNeuro Visor2™ system) may be used in tandem with the Brainsonix ultrasound device to track a patient's brain in virtual space as well as their physical location, thereby ensuring accurate placement.

SUMMARY:
The purpose of this Phase I open label study is to evaluate longer term tolerability and potential effectiveness of transcranial ultrasound in people with tremor as a results of Parkinson's Disease or Essential Tremor.

DETAILED DESCRIPTION:
This study is designed to evaluate the safety and efficacy of focused ultrasound in patients with Parkinson's Disease or Essential Tremor characterized by tremor. The safety of this protocol will be closely monitored and data will be used to determine whether any significant safety issues exist when using focused ultrasound. Adverse events will be noted whenever they occur but will be recorded at the time of the procedure and throughout routine follow-ups, which will persist weekly throughout the duration of the active study protocol. Patients deemed potentially appropriate candidates for focused ultrasound therapy will be treated with 8 sessions of transcranial ultrasound, each of which consists of 10 to 30 minutes of active administration. Clinical and safety outcome measures will be obtained throughout and after completion of the study protocol.

ELIGIBILITY:
Inclusion Criteria:

In order for a subject to be considered for the Essential Tremor application of this study, the following criteria are required:

Subjective complaint of tremor assessed and validated by physician

Must be willing to comply with the study protocol

English Proficiency

At least 18 years of age

At most 90 years of age

In order for a subject to be considered for the Parkinson's Disease application of this study, the following criteria are required:

Diagnosis of Parkinson's Disease validated by physician

Must be willing to comply with the study protocol

English Proficiency

At least 18 years of age

At most 90 years of age

Exclusion Criteria:

In order for a subject to be considered for this study, he/she may NOT have any of the following:

Subjects not English proficient

Subjects unable to give informed consent

Subjects do not meet age requirements (18-90)

Subjects who would not be able to lay down without excessive movement in a calm environment sufficiently long enough to be able to achieve sleep

Pregnancy, women who may become pregnant or are breastfeeding

Women with child-bearing potential who are not willing to use a double-barrier birth control method

Males not willing to use a double-barrier birth control method with female sex partners with child-bearing potential

Advanced terminal illness

Any active cancer or chemotherapy

Any other neoplastic illness or illness characterized by neovascularity

Macular degeneration

Subjects with scalp rash or open wounds on the scalp (for example from treatment of squamous cell cancer)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2024-07-13 (Estimated); Study Completion 2024-08-13 (Estimated)

PRIMARY OUTCOMES:
Essential Tremor Rating Assessment Scale (TETRAS) | Baseline
  The Essential Tremor Rating Assessment Scale was developed by the Tremor Research Group to quantify essential tremor severity and its impact on activities of daily living.
  The ADL section of TETRAS has 12 items, each rated 0, 1, 2, 3 or 4. The maximum total score is 48. Item 1 addresses speech; item 10 addresses occupational impairment; and item 12 assesses social impact. The other 9 items assess activities that are affected primarily by upperweighting of lower limb tremor in the total performance score.
Essential Tremor Rating Assessment Scale (TETRAS) | Through Completion of Study (Average time 8-weeks)
  The Essential Tremor Rating Assessment Scale was developed by the Tremor Research Group to quantify essential tremor severity and its impact on activities of daily living.
  The ADL section of TETRAS has 12 items, each rated 0, 1, 2, 3 or 4. The maximum total score is 48. Item 1 addresses speech; item 10 addresses occupational impairment; and item 12 assesses social impact. The other 9 items assess activities that are affected primarily by upperweighting of lower limb tremor in the total performance score.

SECONDARY OUTCOMES:
9 Hole Pegboard Task (9 HPT) | Baseline
  A validated assessment for fine motor skills, the 9-HPT involves having a participant move 9 pegs individually from starting position to 9 separate peg-holes, as quickly as possible, and to immediately return the 9 pegs to the starting position upon filling the final peg-hole. This is performed separately for each hand. The score is the time (seconds/milliseconds) that it takes to complete the task, recorded separately for dominant and non-dominant hands. The minimum detectable change is 2.6 seconds for the dominant hand and 1.3 seconds for the non-dominant hand.
9 Hole Pegboard Task (9 HPT) | Through Completion of Study (Average time 8-weeks)
  A validated assessment for fine motor skills, the 9-HPT involves having a participant move 9 pegs individually from starting position to 9 separate peg-holes, as quickly as possible, and to immediately return the 9 pegs to the starting position upon filling the final peg-hole. This is performed separately for each hand. The score is the time (seconds/milliseconds) that it takes to complete the task, recorded separately for dominant and non-dominant hands. The minimum detectable change is 2.6 seconds for the dominant hand and 1.3 seconds for the non-dominant hand.
Parkinson's Activities of Daily Living Scale (PAD-L) | Baseline
  The Parkinson's Activities of Daily Living Scale is a self-report activities of daily living scale designed to assess difficulties in daily activities due to symptoms of Parkinson's Disease.
Parkinson's Activities of Daily Living Scale (PAD-L) | Through Completion of Study (Average time 8-weeks)
  The Parkinson's Activities of Daily Living Scale is a self-report activities of daily living scale designed to assess difficulties in daily activities due to symptoms of Parkinson's Disease.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Jordan, MD, Principal Investigator — The Regenesis Project
Locations (1):
- Neurological Associates of West Los Angeles, Los Angeles, California, United States